CLINICAL TRIAL: NCT05770609
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel, Dose-finding Phase II Clinical Study to Evaluate the Efficacy and Safety of SPH3127 Tablets in the Treatment of Mild to Moderate Ulcerative Colitis
Brief Title: A Study of SPH3127 in the Treatment of Mild to Moderate Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPH3127-203
Record Dates: First submitted 2023-03-05; First posted 2023-03-15 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-04

CONDITIONS: Mild to Moderate Ulcerative Colitis
MeSH Terms: interventions — SPH3127

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SPH3127 Tablets with Dose A (Experimental): Oral daily dose of SPH3127 Tablets for up to 8 weeks
  Interventions: Drug: SPH3127 Tablets with Dose A
- SPH3127 Tablets with Dose B (Experimental): Oral daily dose of SPH3127 Tablets for up to 8 weeks
  Interventions: Drug: SPH3127 Tablets with Dose B
- SPH3127 Tablets placebo (Placebo Comparator): Oral daily dose of SPH3127 Tablets placebo for up to 8 weeks
  Interventions: Drug: SPH3127 Tablets placebo

INTERVENTIONS:
Drug: SPH3127 Tablets with Dose A — See Arm description
  Arms: SPH3127 Tablets with Dose A
Drug: SPH3127 Tablets with Dose B — See Arm description
  Arms: SPH3127 Tablets with Dose B
Drug: SPH3127 Tablets placebo — See Arm description
  Arms: SPH3127 Tablets placebo

SUMMARY:
To preliminarily evaluate the clinical efficacy of the renin inhibitor SPH3127 Tablets in patients with mild to moderate ulcerative colitis with placebo as a control and determine the recommended dose.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 - 75 years, male or female;
2. Subjects who have been diagnosed with ulcerative colitis；
3. Subjects who agree to take effective contraceptive measures with their spouses throughout the study period and for up to 12 weeks after the last dose;
4. Subjects who thoroughly learn about the nature, significance, possible benefits, possible inconvenience and potential risks of the trial, understand the study procedures and voluntarily sign the informed consent form prior to their participation in the trial.

Exclusion Criteria:

1. Subjects who are diagnosed with Crohn's disease or indeterminate colitis;
2. Subjects with active infections at screening which may, as evaluated by the investigator, cause increased risks for subjects;
3. Subjects who had surgery that might impact the absorption of oral drugs, subjects who will undergo surgery during the study period, subjects who have undergone major surgery before screening, or subjects who have a plan of surgery during the study period;
4. Subjects and lactating women and those who will become pregnant within 6 months after the trial starts;
5. Subjects with a history of drug abuse with clinical significance within 1 year prior to screening;
6. Subjects with other diseases or conditions that the investigator considers unsuitable for this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Symptom remission rate | Week8
  Symptom remission rate
Endoscopic remission rate | Week8
  Endoscopic remission rate

SECONDARY OUTCOMES:
Clinical remission rate | Week8
  Clinical remission rate
Symptom remission rate | Week2、Week4
  Symptom remission rate
Safety and tolerability since the start of any study treatment. | Approximately 3 months
  Incidence of adverse event and serious adverse event
  , correlation with study drug

CONTACTS AND LOCATIONS:
Locations (25):
- China (25):
  - The First Affiliated Hospital，Sun Yat-sen University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Huizhou First Hospital, Huizhou, Guangdong
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guanmgdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, He'nan
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Henan University, Kaifeng, Henan
  - Union Hospital Tongji Medical College Huazhong Universitu of Science and Technology, Wuhan, Hubei
  - Tongji Hospital Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The First Hospital of Hunan University of Chinese Medicine, Changsha, Hunan
  - The First Affiliated Hospital of University of South China, Hengyang, Hunan
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Shengjing Hospital affiliated to China Medical University, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Xi'an Central Hospital, Xi’an, Shanxi
  - Suining Central Hospital, Suining, Sichuan
  - Beijing Chao-Yang Hospital,Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Chifeng Municipal Hospital, Chifeng
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Shanghai Jiaotong University School of Medicine, Renji Hospital, Shanghai
  - Tianjin Medical University General Hospital;, Tianjin